CLINICAL TRIAL: NCT07076420
Title: Corneal Incision Healing and Its Influencing Factors After Cataract Phacoemulsification in Diabetic Patients -- Based on Anterior Segment Optical Coherence Tomography
Brief Title: Healing of Corneal Incision After Cataract Surgery in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20250122
Record Dates: First submitted 2025-07-14; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Diabetes; Cataract
MeSH Terms: conditions — Diabetes Mellitus; Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Diabetes group
- Control group

SUMMARY:
The objective of this observational study was to understand the healing of corneal incision after cataract surgery in diabetic patients and its influencing factors. The main questions it aims to answer are:

Is corneal incision healing worse in diabetic patients after cataract surgery than in non-diabetic patients? What are the factors affecting corneal incision healing after cataract surgery in diabetic patients?

The results of anterior segment optical coherence tomography before and after cataract surgery in cataract patients with or without diabetes will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

Patients who experience blurred vision and painless visual acuity decline, and are diagnosed with cataract (with or without diabetes) through reliable intraocular pressure, visual acuity and slit lamp examinations, and for whom phacoemulsification of cataract can be considered.

Exclusion Criteria:

* Use multiple eye drops before surgery.
* Complicated by other eye diseases that affect corneal healing, such as keratitis, uveitis, glaucoma, etc.
* Moderate to severe dry eye.
* History of eye surgery.
* Moderate to severe dry eye.
* Grade 5 nuclear cataract.
* Severe systemic diseases (such as chronic renal failure requiring dialysis, severe neurological diseases, immune diseases), pregnancy or lactation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were initially diagnosed with cataract and treated with phacoemulsification and intraocular lens implantation at Zhongnan Hospital of Wuhan University from April 1, 2024 to December 31, 2024.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-15 (Actual)

PRIMARY OUTCOMES:
volume of half cornea with surgical incision | Before surgery; 1 week after surgery; 1 month after surgery
Defect of corneal incision healing | 1 week after surgery; 1 month after surgery
  Opening of internal orifice; Endothelial dislocation; Descemet's membrane detachment

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No